CLINICAL TRIAL: NCT04849377
Title: RBD-HPV: Risk-Based De-Intensification for HPV+ HNSCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of eligible participants due to change in study criterias
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Marshall Posner, MD, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 21-0525
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Human Papillomavirus (HPV); Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Loco Regional Control (LRC); Risk-based De-intensified chemoradio therapy (CRT)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Neoadjuvant Therapy; Carboplatin

STUDY DESIGN:
Intervention Model Description: CRT (Cisplatin with IMRT/IMPT): Group I 50 Gy/200 mg/m2, Group II 54 Gy/200 mg/m2, Group III 60 Gy/240 mg/m2 Sequential Therapy: Group IV TPF Induction followed by 60 Gy and Carboplatin AUC 1.5
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I - 50 Gy/200 mg/m2 (Experimental): Patient Characteristics: <20 Pack-Years, HPV16, OP, T1,T2 N0 RT 5 days per week for 6 weeks and Cisplatin weekly for 5 weeks
  Interventions: Radiation: RT 50 Gy; Drug: Cisplatin 200
- Group II - 54 Gy/200mg/m2 (Experimental): Patient Characteristics: <20 Pack-Years, HPV16, OP, T1-T2, N1-N2b, T3 N0-N2b RT 5 days per week for 6 weeks and Cisplatin weekly for 6 weeks
  Interventions: Radiation: RT 54 GY; Drug: Cisplatin 200
- Group III - 60 Gy/240 mg/m2 (Experimental): Patient Characteristics: 20-40 Pack-Years, Non-HPV16, Non-OP, T1-T2, N1-N2b, T3 N0-N2b RT 5 days per week for 6 weeks and Cisplatin weekly for 6 weeks
  Interventions: Radiation: RT 60 GY; Drug: Cisplatin 240
- Group IV - TPF Induction followed by 60 Gy and Carboplatin AUC 1.5 (Experimental): Patient Characteristics: 20-40 Pack-Years, Non-HPV16, Non-OP, T4, N2c, >3 nodes, ENE, or Matted Nodes Induction Therapy: Cisplatin, Docetaxel, Fluorouracil followed by RT 60 GY + Carboplatin AUC 9.0 Docetaxel every 21 days for 3 cycles, Cisplatin every 21 days for 3 cycles, Fluorouracil continuous infusion over 4 days (every 21 days for 3 cycles). Followed by RT 5 days per week for 6 weeks and Carboplatin weekly for 6 weeks.
  Interventions: Radiation: RT 60 GY; Other: Induction Therapy; Drug: Carboplatin; Drug: Cisplatin 240

INTERVENTIONS:
Radiation: RT 50 Gy — Radiation Therapy (RT) 50 GY
  Other Names: Radiation Therapy
  Arms: Group I - 50 Gy/200 mg/m2
Radiation: RT 54 GY — Radiation Therapy (RT) 54 GY
  Other Names: Radiation Therapy
  Arms: Group II - 54 Gy/200mg/m2
Radiation: RT 60 GY — Radiation Therapy (RT) 60 GY
  Other Names: Radiation Therapy
  Arms: Group III - 60 Gy/240 mg/m2; Group IV - TPF Induction followed by 60 Gy and Carboplatin AUC 1.5
Other: Induction Therapy — Induction Therapy: Cisplatin, Docetaxel, Fluorouracil
  Arms: Group IV - TPF Induction followed by 60 Gy and Carboplatin AUC 1.5
Drug: Carboplatin — Carboplatin AUC 9.0
  Arms: Group IV - TPF Induction followed by 60 Gy and Carboplatin AUC 1.5
Drug: Cisplatin 200 — 200 mg/m2
  Arms: Group I - 50 Gy/200 mg/m2; Group II - 54 Gy/200mg/m2
Drug: Cisplatin 240 — 240mg/m2
  Arms: Group III - 60 Gy/240 mg/m2; Group IV - TPF Induction followed by 60 Gy and Carboplatin AUC 1.5

SUMMARY:
The purpose of this research study is to determine the rate of local regional control at 2 years when using de-intensified chemoradiotherapy (CRT) in patients with Human Papillomavirus (HPV)-associated head and neck squamous cell carcinoma (HNSCC). Local regional control means no recurrence of the cancer in the head or neck area. Study subjects will be enrolled into 4 groups. Group/treatment will be based on a number of factors, including smoking and drinking history.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the rate of local regional control at 2 years when using de-intensified chemoradiotherapy (CRT) in patients with Human Papillomavirus (HPV)-associated head and neck squamous cell carcinoma (HNSCC). Local regional control means no recurrence of the cancer in the head or neck area. Study subjects will be enrolled into 4 groups. Group/treatment will be based on a number of factors, including smoking and drinking history.

If participants choose to participate, participants will be asked to:

* Participate in screening for eligibility, this will include: questions regarding \medical history, physical exam, blood/urine samples, electrocardiogram, PET/CT and/or CT-MRI of the neck, assessment of tumor, and a questionnaire.
* Complete the study regimen including evaluations and follow up visits. Participants may be in this research study for approximately to 5 years after receiving standard of care (SOC) treatment. Depending on the group enrolled in, the treatment will last either 6 weeks (Groups 1-3) or 15 weeks (Group 4.This group will also receive 3 cycles of SOC induction therapy (One cycle = 21 days). Induction therapy is initial chemotherapy delivered prior to radiation or surgery when treating cancer.
* Participate in routine types of procedures such as clinical exams, blood and urine tests, and imaging tests to assess tumor.
* Consent to storage of research samples.

This research study involves chemotherapy and intensity-modulated radiation therapy (IMRT) IMRT is used to safely deliver precise radiation to a tumor while minimizing the dose to surrounding normal tissue.

There are no added costs associated with participation. There is no reimbursement for participation.

The names of the drugs/interventions involved in this study are:

* Cisplatin
* Docetaxel (Group 4 only)
* Fluorouracil (Group 4 only)
* Carboplatin (Group 4 Only)

All of the drugs listed above are approved for use by the Food and Drug Administration (FDA), commercially available, and considered standard of care (SOC) for cancer.

Serious known side effects that participants may experience include:

* Nausea and vomiting
* Diarrhea
* Fever
* Skin irritation, rash
* Joint pain

ELIGIBILITY:
Inclusion Criteria: Patients must meet the following inclusion criteria to be eligible for enrollment in RBD-HPV:

1. Histologically-confirmed squamous cell carcinoma of the head and neck, including subsites of the oropharynx, hypopharynx, larynx, and nasopharynx (with data on EBV)
2. P16+ positivity as measured by IHC in a lab that is verified by the central laboratory or if the slides are available for review by the central laboratory
3. HPV positivity by PCR assessed with either tissue or cytology in the central laboratory
4. Stages I, II, III, or IV according to the AJCC 7th edition without evidence of distant metastases
5. Age > 18
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Adequate marrow function as defined by the following parameters:

   * Neutrophil count > 1.5 x 109/l
   * Platelet count > 100 x 109/l
   * Hemoglobin > 10 g/dl
8. Adequate renal function as defined by a creatinine clearance > 60 ml/min (actual or calculated by the Cockcroft-Gault equation)
9. Adequate liver function as defined by the following parameters:

   * Total bilirubin < institutional upper limit of normal (ULN) (except patients with Gilbert's Syndrome who have no other liver disease or abnormal liver serologies)
   * AST or ALT and alkaline phosphatase within the ranges described below
10. A negative pregnancy test within 7 days of starting therapy in women of childbearing potential
11. Capacity to understand the study protocol
12. Willingness to provide written consent.

Exclusion Criteria: Patients will not be eligible for enrollment in this study if they exhibit any of the following conditions:

1. Women who are currently pregnant or breast-feeding
2. Men or women of childbearing potential who are not using adequate contraception during treatment and at least 3 months after therapy
3. Current or prior malignancy in the last 5 years (excluding basal or squamous cell carcinoma of the skin not requiring systemic or radiation therapies, or prostate CA that is well-controlled and observed, etc)
4. Radiation therapy for prior malignancy (except radioactive iodine for thyroid cancer)
5. Prior chemotherapy for other malignancy or autoimmune disease
6. Metastatic disease at presentation
7. Nasal cavity subsite
8. Active smoking (defined as > 1 cigarette per day within the last five years) or former smoking (has to have quit > 10 years ago) with a cumulative pack year history > 40 pack years
9. Prior radiation therapy or chemotherapy for HNSCC (prior surgery alone is permitted)
10. Active substance use disorder (ETOH or drugs, excluding marijuana)
11. Prior use of IV drugs
12. Significant peripheral neuropathy (> grade 2 according to NCI CTC)
13. Prior hematologic or solid organ transplant
14. Major medical comorbidity including:

    * Significant cardiovascular disease.
    * Significant neurologic disorder, including dementia and seizures.
    * Significant psychiatric disorder.
    * Active infection that is uncontrolled.
    * PUD (peptic ulcer disease) that is clinically active or unhealed.
    * Hypercalcemia.
    * COPD with hospitalization in the last 12 months for pneumonia or respiratory failure.
    * Interstitial lung disease.
    * Autoimmune disease requiring therapy.
    * Uncontrolled HIV infection (not on HAART, CD4 < 200).
    * Active Hepatitis C (+ RNA).
15. Enrollment in a therapeutic clinical trial within 30 days of study entry
16. Concurrent treatment with any other antineoplastic therapy
17. Significant weight loss (> 25% of TBW) in the 2 months prior to study entry
18. Patient has a history of non-adherence to medical care
19. Patient will not be able to engage in comprehensive follow-up at Mount Sinai.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Rate of Locoregional control (LRC) | 2 years
  The rate of locoregional control (LRC) at 2 years - Local regional control means no recurrence of the cancer in the head or neck area.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Principal Investigator — Ichan School of Medicine at Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
All of the individual participant data collected during the trial, after deidentification.

REFERENCES:
- [Background] D'Souza G, Kreimer AR, Viscidi R, Pawlita M, Fakhry C, Koch WM, Westra WH, Gillison ML. Case-control study of human papillomavirus and oropharyngeal cancer. N Engl J Med. 2007 May 10;356(19):1944-56. doi: 10.1056/NEJMoa065497. PMID 17494927
- [Background] Carlander AF, Gronhoj Larsen C, Jensen DH, Garnaes E, Kiss K, Andersen L, Olsen CH, Franzmann M, Hogdall E, Kjaer SK, Norrild B, Specht L, Andersen E, van Overeem Hansen T, Nielsen FC, von Buchwald C. Continuing rise in oropharyngeal cancer in a high HPV prevalence area: A Danish population-based study from 2011 to 2014. Eur J Cancer. 2017 Jan;70:75-82. doi: 10.1016/j.ejca.2016.10.015. Epub 2016 Nov 23. PMID 27888679
- [Background] Klussmann JP, Mooren JJ, Lehnen M, Claessen SM, Stenner M, Huebbers CU, Weissenborn SJ, Wedemeyer I, Preuss SF, Straetmans JM, Manni JJ, Hopman AH, Speel EJ. Genetic signatures of HPV-related and unrelated oropharyngeal carcinoma and their prognostic implications. Clin Cancer Res. 2009 Mar 1;15(5):1779-86. doi: 10.1158/1078-0432.CCR-08-1463. Epub 2009 Feb 17. PMID 19223504
- [Background] Mork J, Lie AK, Glattre E, Hallmans G, Jellum E, Koskela P, Moller B, Pukkala E, Schiller JT, Youngman L, Lehtinen M, Dillner J. Human papillomavirus infection as a risk factor for squamous-cell carcinoma of the head and neck. N Engl J Med. 2001 Apr 12;344(15):1125-31. doi: 10.1056/NEJM200104123441503. PMID 11297703
- [Background] Seiwert TY, Zuo Z, Keck MK, Khattri A, Pedamallu CS, Stricker T, Brown C, Pugh TJ, Stojanov P, Cho J, Lawrence MS, Getz G, Bragelmann J, DeBoer R, Weichselbaum RR, Langerman A, Portugal L, Blair E, Stenson K, Lingen MW, Cohen EE, Vokes EE, White KP, Hammerman PS. Integrative and comparative genomic analysis of HPV-positive and HPV-negative head and neck squamous cell carcinomas. Clin Cancer Res. 2015 Feb 1;21(3):632-41. doi: 10.1158/1078-0432.CCR-13-3310. Epub 2014 Jul 23. PMID 25056374
- [Background] Gillison ML, D'Souza G, Westra W, Sugar E, Xiao W, Begum S, Viscidi R. Distinct risk factor profiles for human papillomavirus type 16-positive and human papillomavirus type 16-negative head and neck cancers. J Natl Cancer Inst. 2008 Mar 19;100(6):407-20. doi: 10.1093/jnci/djn025. Epub 2008 Mar 11. PMID 18334711
- [Background] Gillison ML, Chaturvedi AK, Anderson WF, Fakhry C. Epidemiology of Human Papillomavirus-Positive Head and Neck Squamous Cell Carcinoma. J Clin Oncol. 2015 Oct 10;33(29):3235-42. doi: 10.1200/JCO.2015.61.6995. Epub 2015 Sep 8. PMID 26351338
- [Background] Marur S, D'Souza G, Westra WH, Forastiere AA. HPV-associated head and neck cancer: a virus-related cancer epidemic. Lancet Oncol. 2010 Aug;11(8):781-9. doi: 10.1016/S1470-2045(10)70017-6. Epub 2010 May 5. PMID 20451455
- [Background] Dayyani F, Etzel CJ, Liu M, Ho CH, Lippman SM, Tsao AS. Meta-analysis of the impact of human papillomavirus (HPV) on cancer risk and overall survival in head and neck squamous cell carcinomas (HNSCC). Head Neck Oncol. 2010 Jun 29;2:15. doi: 10.1186/1758-3284-2-15. PMID 20587061
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Westra WH, Taube JM, Poeta ML, Begum S, Sidransky D, Koch WM. Inverse relationship between human papillomavirus-16 infection and disruptive p53 gene mutations in squamous cell carcinoma of the head and neck. Clin Cancer Res. 2008 Jan 15;14(2):366-9. doi: 10.1158/1078-0432.CCR-07-1402. PMID 18223210
- [Background] Fakhry C, Westra WH, Li S, Cmelak A, Ridge JA, Pinto H, Forastiere A, Gillison ML. Improved survival of patients with human papillomavirus-positive head and neck squamous cell carcinoma in a prospective clinical trial. J Natl Cancer Inst. 2008 Feb 20;100(4):261-9. doi: 10.1093/jnci/djn011. Epub 2008 Feb 12. PMID 18270337
- [Background] Chaturvedi AK, Anderson WF, Lortet-Tieulent J, Curado MP, Ferlay J, Franceschi S, Rosenberg PS, Bray F, Gillison ML. Worldwide trends in incidence rates for oral cavity and oropharyngeal cancers. J Clin Oncol. 2013 Dec 20;31(36):4550-9. doi: 10.1200/JCO.2013.50.3870. Epub 2013 Nov 18. PMID 24248688
- [Background] Braakhuis BJ, Snijders PJ, Keune WJ, Meijer CJ, Ruijter-Schippers HJ, Leemans CR, Brakenhoff RH. Genetic patterns in head and neck cancers that contain or lack transcriptionally active human papillomavirus. J Natl Cancer Inst. 2004 Jul 7;96(13):998-1006. doi: 10.1093/jnci/djh183. PMID 15240783
- [Background] Lassen P, Eriksen JG, Hamilton-Dutoit S, Tramm T, Alsner J, Overgaard J. Effect of HPV-associated p16INK4A expression on response to radiotherapy and survival in squamous cell carcinoma of the head and neck. J Clin Oncol. 2009 Apr 20;27(12):1992-8. doi: 10.1200/JCO.2008.20.2853. Epub 2009 Mar 16. PMID 19289615